CLINICAL TRIAL: NCT02668835
Title: GADGET-PD Genetic and Digital Diagnosis of Essential Tremor and Parkinson's Disease Trial
Acronym: GADGET-PD
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Intel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-15-6628
Record Dates: First submitted 2015-12-04; First posted 2016-01-29 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Idiopathic Parkinson's Disease as defined by the UK brain bank criteria and history of resting tremor.
  Interventions: Device: Non intervention-Monitoring device; Genetic: Non intervention-Genetic testing
- Cohort 2: Essential Tremor with history of resting tremor. Diagnosis made by a movement disorder specialist
  Interventions: Device: Non intervention-Monitoring device; Genetic: Non intervention-Genetic testing

INTERVENTIONS:
Device: Non intervention-Monitoring device — Fox Insight self-monitoring android app and smartwatch Participants will be asked to wear a smartwatch with accelerometers, during day and night, for a period of 2 weeks. Additionally, a self-monitoring app on a smartphone is used, where the participant reports when they take any medication and performs a focused attention task to encourage resting tremor.
Genetic: Non intervention-Genetic testing

SUMMARY:
The proposed study will capitalize on the early predictive information stored in an individual's genetic risk for Parkinson Disease (PD) in combination with the subtle features of tremors that can be extracted from movement data gathered by modern compact accelerometers in order to determine if accurate discrimination of essential tremor (ET) from PD can be achieved. Both of these technologies have a proven but somewhat limited ability to inform diagnosis of PD or differentiation of PD from ET - especially at early stages of the disease. The investigators hypothesize that a combination of prior genetic risk and current disease symptomology can synergize for accurate and early discrimination of PD from ET and ultimately inform a cost effective approach to movement disorder diagnosis.

In this study, the investigators will collect blood from individuals with confirmed late-onset diagnosis of PD and ET. Gold standard diagnosis status will be determined via the Unified Parkinson's Disease Rating Scale (UPDRS) - the accepted clinical gold standard for Parkinson's Disease diagnosis. DNA will be extracted from blood samples to characterize the genetic risk of individuals for PD via proven genetic risk models. In addition, participants will wear a wristwatch-like accelerometer device that will track their movements (tremors) at high temporal resolution and transmit movement data via a smartphone. Cognitive distraction tasks will be administered via mobile phones while simultaneously collecting movement data. Predictive tremor features will be extracted from movement data via signal processing approaches - e.g. discrete wavelet transformation. A final predictive model combining movement tracking information and genetic information will be designed in attempt to distinguish PD from ET individuals.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease as defined by the UK brain bank criteria and history of resting tremor, or:
* Essential Tremor with history of resting tremor. Diagnosis made by a movement disorder specialist.
* Midstage in disease process for Parkinson's disease with history of resting tremor

Exclusion Criteria:

* Dementia as defined by a mini-mental state examination cutoff score of 27
* Atypical Parkinsonism
* Akinesia/ rigidity Parkinson's Disease
* Movement Disorders - Stiff-Person syndrome, choreatic disease, dystonia, progressive supranuclear palsy
* Motor neuron disease - Multiple sclerosis, amyotrophic lateral sclerosis, motor neuritis, progressive bulbar palsy, progressive muscular atrophy, spinal muscular atrophy
* Significant neurological comorbidities:

  * Stroke
  * Brain cancer or brain metastases
* History of bone marrow transplant
* Cerebral palsy and spastic paraplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is limited to individuals presenting in Scripps Health clinics with diagnosis of Parkinson's disease or essential tremor.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Comparison of genetic markers between cohorts (Parkinson's disease and Essential Tremor) | 2 years
  The primary outcome of the study is the generation of genomic information that may inform the diagnosis and/or treatment of movement disorders. The endpoint will be derived from the successful implementation of genomic assays, appropriate bioinformatic and statistical analysis of the genomic data generated by those assays. These analyses and report generation activity may be based on comparison of the genomic profile of a patient with data obtained from other such studies or publicly available data in addition to comparison between datasets generated within this study.
Tremor frequency over two week period | 2 weeks
  A primary outcome of the study is the tremor frequency over two week period that may inform the diagnosis and/or treatment of movement disorders. The endpoint will be derived data recorded from a digital wristwatch-like device. These analyses and report generation activity may be based on comparison between datasets generated within this study.

SECONDARY OUTCOMES:
Comparison of genetic markers to tremor characteristics | 2 years
  Secondary outcomes for this analysis include the identification of genetic characteristics that differentiate individuals with specific tremor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Torkamani, PhD, Principal Investigator — Scripps Translational Science Institute